CLINICAL TRIAL: NCT02110108
Title: Study for the RevLite Laser System for Facial Solar Lentigines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN14-REV-REJUV-NS
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Facial Solar Lentigines

STUDY DESIGN:
Intervention Model Description: Each patient receives a single wavelength treatment on one side of their face, and a double wavelength on the other side of their face.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Revlite Laser System- Single Wavelength (Experimental): Revlite Laser System- 1064nm wavelength will be used on half of the face.
  Interventions: Device: Revlite Laser System
- Revlite Laser System- Dual Wavelength (Experimental): Revlite Laser System- treatment will consist of 1064 nm and 532 nm wavelengths on half of the face.
  Interventions: Device: Revlite Laser System

INTERVENTIONS:
Device: Revlite Laser System — Revlite Laser System for the Treatment of Facial Solar Lentigines

SUMMARY:
The purpose of this study is to evaluate the effects of the Revlite Laser System for treatment of facial solar lentigines

DETAILED DESCRIPTION:
Prospective facial study using the revlite laser to treat pigmentation caused by sun damage.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 60 years old.
2. Is Fitzpatrick Skin types I-III
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.
5. Has clinically determined mild to severe facial mottled pigmentation (solar lentigines) on the face.

Exclusion Criteria:

1. Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. Is hypersensitive to light exposure OR takes photo sensitized medication.
3. Has active or localized systemic infections.
4. Has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to the heavy use of aspirin {greater than 81 mg per day}).
5. Has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. Is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. Has used Accutane within 6 months prior to enrollment.
8. Has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. Has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. Has a history of keloids.
11. Has evidence of compromised wound healing.
12. Has a history of basal cell carcinoma, squamous cell carcinoma or melanoma.
13. Has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications or has an autoimmune disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Sadick Research Group, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Revlite Laser System: Revlite Laser System
  Revlite Laser System: Revlite Laser System with ½ of the face treated with the 1064nm wavelength and the other half of the face treated with combination of both the 1064nm and 532nm wavelengths.
Period: Overall Study
Arm/Group | Revlite Laser System
Started | 10
RevLite Single Wavelength | 10
RevLite Combo Wavelength | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Revlite Laser System: Revlite Laser System
  Revlite Laser System: Revlite Laser System for the Treatment of Facial Solar Lentigines
Arm/Group | Revlite Laser System
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 8
  Race/Ethnicity: Hispanic | 2
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 1
    Fitzpatrick Skin Type II | 7
    Fitzpatrick Skin Type III | 2
    Fitzpatrick Skin Type IV | 0
    Fitzpatrick Skin Type V | 0
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Photographic Evaluation Using the Blinded Global Aesthetic Improvement Scale
Description: Photos taken at baseline will be compared to photos taken 1 month post last treatment to assess the level of improvement using the Global Aesthetic Improvement Scale. This evaluation is blinded. This scale ranges from -1 to 3, where -1 is worsened, 0 is no change, 1 is improved, 2 is much improved, and 3 is very much improved.
Time Frame: 1 month post last treatment
Population: Since all subjects who enrolled received at least 1 treatment and had a 30 day follow up to this treatment, all subject information is included. The time frame is based off of the follow up to each subject's final treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Revlite Laser System Single: Revlite Laser System using just 1064 nm wavelength
- Revlite Laser System- Combo: Revlite Laser System using 1064 nm and 532 nm wavelengths
Arm/Group | Revlite Laser System Single | Revlite Laser System- Combo
Number analyzed (Participants) | 10 | 10
Participants
  Very Much Improved | 0 | 1
  Much Improved | 3 | 3
  Improved | 6 | 4
  No Change | 1 | 2
  Worse | 0 | 0

2. Secondary Outcome: Physician Satisfaction Questionnaire
Description: The satisfaction is on a scale ranging from extremely satisfied (6) to extremely dissatisfied (1).
Time Frame: 1 month post last treatment
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- Revlite Laser System- Single: Revlite Laser System with just 1064 nm wavelength used.
- Revlite Laser System- Combo: Revlite Laser System with both 1064 nm and 532 nm used.
Arm/Group | Revlite Laser System- Single | Revlite Laser System- Combo
Number analyzed (Participants) | 10 | 10
score on a scale | 3.70 (1.63) | 3.600 (1.65)

ADVERSE EVENTS:
Time Frame: Adverse events occurring will be captured and followed throughout each subject's participation in the study, approximately 8 months.
Groups:
- Revlite Laser System Single: Revlite Laser System
  Revlite Laser System 1064nm wavelength
- Revlite Laser System Combo: Revlite Laser System
  Revlite Laser System: Combination of both the 1064nm and 532nm wavelengths
Arm/Group | Revlite Laser System Single | Revlite Laser System Combo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Revlite Laser System Single (N=10) | Revlite Laser System Combo (N=10)
Pain (Nervous system disorders) | 5 | 5
Redness (Skin and subcutaneous tissue disorders) | 9 | 9
Swelling (Skin and subcutaneous tissue disorders) | 5 | 3
Crusting (Skin and subcutaneous tissue disorders) | 4 | 4
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.